CLINICAL TRIAL: NCT00470418
Title: Development of NIC5-15 in the Treatment of Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Humanetics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MHBB-009-06S; R21AT003302-01A1 (NIH)
Record Dates: First submitted 2007-05-04; First posted 2007-05-07 (Estimated); Results first posted 2017-01-09 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Alzheimer Disease; Dementia
Keywords: Alzheimer Disease; Alzheimer Type Senile Dementia; Alzheimer's Disease; clinical trial; dementia; diabetes; dietary supplements; Senile Dementia, Alzheimer Type; Therapeutics
MeSH Terms: conditions — Alzheimer Disease; Dementia; Diabetes Mellitus | interventions — pinitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NIC5-15 (Other): Subjects with Alzheimer's Disease
  Interventions: Drug: NIC5-15
- Placebo (Placebo Comparator): Subjects with Alzheimer's Disease
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NIC5-15 — a natural product, found in many foods and plants with mild insulin sensitizing effects
  Other Names: d-Pinitol
  Arms: NIC5-15
Drug: Placebo — placebo comparator
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of NIC5-15in the treatment of Alzheimer's Disease.

DETAILED DESCRIPTION:
Recent epidemiologic evidence, has suggested that diabetes mellitus significantly increases risk for the development of Alzheimer's disease, independent of vascular risk factors. Moreover, even patients who are simply insulin resistant, without frank diabetes, have been shown to share this elevated risk for the development of AD. As insulin's role as a neuromodulator in the brain has been revealed, several potential mechanisms for the interaction of diabetes or insulin resistance with AD have been suggested such as decreased cortical glucose utilization particularly in the hippocampus and entorhinal cortex; increased oxidative stress through the formation of advanced glycation end products; increased Tau phosphorylation and neurofibrillary tangle formation; and increased beta-amyloid aggregation through inhibition of insulin-degrading enzyme. The future treatment of AD might involve pharmacologic and dietary manipulations of insulin and glucose regulation

NIC5-15 is a single, small, naturally occurring molecule. Animal studies and some human trials have shown NIC5-15 to be safe and a potent insulin sensitizer at doses equivalent to 800-2000mg per day. In preclinical studies at doses higher than those previously studied in clinical trials, we found that NIC5-15 interferes with the accumulation of beta amyloid, an important step in the development of Alzheimer's pathology. These data suggest that NIC5-15 may be a reasonable therapeutic agent for the treatment of Alzheimer Disease for two reasons:

1. It is a -secretase inhibitor that is Notch-sparing.
2. It is potentially an insulin-sensitizer.

However critical safety and human efficacy studies must be conducted. This application proposes to conduct these early critical human studies. The goal of the studies contained in this proposal is to establish safety and efficacy of NIC5-15 for the treatment of AD. The specific objectives of this study are to:

Specific Objective #1) Conduct a multiple dose safety study of NIC5-15 to establish safety in the doses that appear to block amyloid accumulation. These studies will characterize the safety profile, pharmacokinetics, and tolerability

Specific Objective #2) Conduct a double blind placebo controlled pilot efficacy study of NIC5-15 in patients with AD. The goals of this study are to:

A) Demonstrate feasibility for a multi-site trial that will be used to guide the design of a future larger effort. Demonstration of feasibility will include examination of accrual rate, overall recruitment, adherence to protocol, compliance with medication and willingness to complete a randomized trial, and lack of short term toxicity.

B) Collect preliminary evidence of efficacy in terms of cognitive and global measures as well as secondary efficacy outcomes of activities of daily living, behavioral disturbances and AD biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* NINCDS/ADRDA criteria for probable AD
* MMSE between 12-27
* Treatment with a cholinesterase inhibitor or an NMDA (N-methyl-D-asparate) antagonist with stable dose for at least 12 weeks
* Home monitoring available for supervision of medications
* Caregiver available to accompany patient to all visits and willing to participate in study as informant
* Fluent in English or Spanish
* Medical stability for this study as confirmed by review of records, internist's physical exam, neurological exam, and laboratory tests
* Stable doses of non-excluded medication
* No evidence of hepatic insufficiency
* Able to swallow oral medications
* Ability to participate in the informed consent process

Exclusion Criteria:

* History of Diabetes Mellitus (OGTT criteria) requiring treatment with an excluded antidiabetic medication (see below) or history of hypoglycemia
* Active hepatic or renal disease
* Cardiac disease including history of congestive heart failure or current treatment for CHF; history of recent myocardial infarction
* Use of another investigational drug within the past two months
* History of clinically significant stroke
* History of seizure or head trauma with disturbance of consciousness within the past two years
* Major mental illness including psychotic disorders, bipolar disorder, or major depressive episode within the past two years Medication Exclusion
* Current use of oral hypoglycemic agents including sulfonylureas and meglintinides
* Current use of a lipid-lowering agent (excluded from Study #1, see discussion below)
* Current or past treatment with insulin for longer than two weeks
* Current use of drugs with significant anticholinergic or antihistaminic properties

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-01; Primary Completion 2008-08 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hillel Grossman, MD, Principal Investigator — VA Medical Center, Bronx
Locations (1):
- VA Medical Center, Bronx, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5 subjects did not meet entry criteria and were not baselined
Groups:
- NIC5-15: NIC5-15: a natural product, found in many foods and plants with mild insulin sensitizing effects. Subjects received escalating doses of 1500, 3000 and 5000 mg daily over the course of the study.
  Subjects with Alzheimer's Disease
- Placebo: Placebo: placebo comparator identical in pill size, appearance and number
  Subjects with Alzheimer's Disease
Period: Overall Study
Arm/Group | NIC5-15 | Placebo
Started | 7 | 3
Completed | 6 | 3
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NIC5-15 | Placebo | Total
Number analyzed (Participants) | 7 | 3 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.4 (12.5) | 69.7 (13.9) | 70.05 (.49)
Gender [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 4 | 2 | 6
Education [Mean (Standard Deviation); unit: Years of Education] | 12.3 (4.6) | 18.0 (2.0) | 15.15 (4.0)

OUTCOME MEASURES:

1. Primary Outcome: Safety Assessments: Number of Participants With Adverse Events
Description: vital signs, physical exam, Symptom Checklist, complete blood count, serum chemistries, urinalysis, and electrocardiogram
Time Frame: Safety Labs, Physical Exams: 6 times over 7 weeks. Adverse Events assessed 21 times over the course of 7 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | NIC5-15 | Placebo
Number analyzed (Participants) | 7 | 3
Participants | 07 | 02

2. Secondary Outcome: Changes From Baseline in Clinical Measures of Cognition at Terminal Visit
Description: Mini-Mental Status Exam (MMSE) 0(worst)-30(best); ADAS-cog 0 (best cognitive performance across multiple domains) - 70(worst); Activities of Daily Living (ADCS-ADL) 0(least capable of function in daily and instrumental activities)-54(best)
Time Frame: baseline and six weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NIC5-15 | Placebo
Number analyzed (Participants) | 7 | 3
units on a scale
  MMSE | .8 (1.02) | -5.3 (6.4)
  ADAS-cog | 2 (2.1) | 5.3 (3.2)
  ADCS-ADLs | 1 (2.8) | 1.7 (7.4)

ADVERSE EVENTS:
Arm/Group | NIC5-15 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/3
Other Adverse Events (participants affected / at risk) | 7/7 | 2/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NIC5-15 (N=7) | Placebo (N=3)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Fall (Social circumstances) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Joint Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vomitting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Scratchy Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hyperglycemic Lab Value (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Discomfort and Pain at Needle Injection Site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Hypoglycemic Lab Value (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Low Hemocrit Lab Value (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Patient had chronic anemia
Bleeding from Scratch on Arm (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No